CLINICAL TRIAL: NCT05816317
Title: A Single-session Intervention for Suicidal Thoughts and Behaviors
Brief Title: Randomized Controlled Trial of a Single-session Mechanism-focused Intervention for Suicidal Thoughts and Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shannon E. Sauer-Zavala (Other)
Responsible Party: Sponsor-Investigator, Shannon E. Sauer-Zavala, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 343205
Record Dates: First submitted 2023-03-29; First posted 2023-04-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation; Hopelessness; Wish to Live; Wish to Die
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Session Mechanism Focused Intervention (SSMFI) (Experimental)
  Interventions: Behavioral: Single-Session Mechanism-Focused Intervention (SSMFI)
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Distress Tolerance Skills Review

INTERVENTIONS:
Behavioral: Single-Session Mechanism-Focused Intervention (SSMFI) — A brief intervention for patients hospitalized for suicide risk that directly targets hopelessness and perceptions of social relatedness.
  Arms: Single-Session Mechanism Focused Intervention (SSMFI)
Behavioral: Distress Tolerance Skills Review — Treatment as usual at the inpatient setting for this study.
  Arms: Treatment as Usual

SUMMARY:
Across multiple models of suicide risk, hopelessness and perceptions of social relatedness (i.e., lack of social connection/thwarted belongingness, perceived burdensomeness) have emerged as candidate mechanisms that maintain STBs. Although these mechanisms have garnered strong empirical support in predicting STBs, there has been virtually no integration with interventions aimed for individuals at acute risk for suicide. Thus, the overarching goal of the present proposal is to evaluate a mechanism-focused intervention that explicitly targets two core mechanisms implicated in the maintenance of STBs: hopelessness and negative perceptions of social relatedness. Given that the period immediately following hospital discharge presents the highest risk for suicide attempts and up to 70% of patients admitted for a suicide attempt do not attend their first outpatient appointment, the intervention will be evaluated on an inpatient unit. Additionally, most of the extant interventions for STBs are administered across multiple sessions (i.e., 4 sessions and up to one year); however treatments of this length are unlikely to be feasible in acute care settings. Fortunately, very brief suicide prevention interventions, are effective in reducing future suicide attempts and increasing the likelihood of attending follow-up treatments. Additionally, single-session interventions (not suicide specific) have been shown to reduce hopelessness immediately and at a one-month follow-up.

The present study is an RCT comparing a novel Single Session Mechanism Focused Intervention (SSMFI) for STBs to treatment-as-usual (TAU) on a psychiatric inpatient unit for patients admitted for suicidal ideation or attempt. The engagement of the putative processes (hopelessness and negative perceptions of social relatedness) that maintain STBs will be assessed, along with the feasibility and acceptability of SSMFI for STBs on an inpatient psychiatric unit.

ELIGIBILITY:
Inclusion Criteria:

* admitted for care to the Adult Inpatient Unit at Good Samaritan Hospital
* endorse suicidal ideation and/or a recent suicide attempt (i.e., "a potentially self-injurious act committed with at least some wish to die") upon intake to the unit
* 18 years of age; (4) English speaking
* able to provide two methods for follow-up contact (i.e., phone number, email address) in order to complete study follow-up assessment.

Exclusion Criteria:

* current manic episode
* acutely psychotic
* actively detoxicating from substances
* the inability to comprehend the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in intensity of suicidal ideation | Pre-intervention and directly after the intervention (i.e., 1 hour later)
  RATE OVERALL INTENSITY OF YOUR SUICIDAL IDEATION RIGHT NOW: (scale from "1" Extremely low intensity to "5" Extremely high intensity)
Change in hopelessness | Pre-intervention and directly after the intervention (i.e., 1 hour later)
  How much are you feeling hopeless right now? (scale from "1" Not at all to "5" A lot)
Change in wish to live | Pre-intervention and directly after the intervention (i.e., 1 hour later)
  I wish to live this much: (scale from "0" Not at all to "8" Very much)
Change in wish to die | Pre-intervention and directly after the intervention (i.e., 1 hour later)
  I wish to die this much: (scale from "0" Not at all to "8" Very much)
Change in Beck Hopelessness Scale | pre-intervention, 1 week after the intervention is completed, 1 month after the intervention is completed
  Hopelessness will be measured with the Beck Hopelessness Scale. Scores range from 0-20 and higher scores indicate greater levels of hopelessness.
Change in Interpersonal Needs Questionnaire | pre-intervention, 1 week after the intervention is completed, 1 month after the intervention is completed
  Perceptions of social connectedness will be assessed with the Interpersonal Needs Questionnaire. Scores range from 0 to 107 with higher scores indicating less connection with others.

SECONDARY OUTCOMES:
Change in Columbia Suicide Severity Rating Scale | pre-intervention, 1 week after the intervention is completed, 1 month after the intervention is completed
  The self-report version of the Columbia Suicide Severity Rating Scale will be used to assess the presence of suicidal behaviors thoughts and behaviors. Participants are asked to respond Yes/No to 6 items that refer to various suicide related phenomena (thoughts, planning, intent, and behaviors). There is no total score for this measure.
Change in Adult Suicidal Ideation Questionnaire | pre-intervention, 1 week after the intervention is completed, 1 month after the intervention is completed
  Intensity of suicidal ideation will be measured with the Adult Suicidal Ideation Questionnaire. Scores range from 0-150 and higher scores indicate greater intensity of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No